CLINICAL TRIAL: NCT03282643
Title: Rivaroxaban Versus Low-molecular-weight Heparin in Preventing Thrombosis Among Cancer Patients After Femoral Venepuncture
Brief Title: Rivaroxaban Versus Low-molecular-weight Heparin for Preventing Thrombosis in Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Dean & Director, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rivaroxaban vs heparin
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Rivaroxaban; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rivaroxaban 10mg daily (Experimental): orally, 10 mg once daily for day1 and day 2 after femoral venepuncture
  Interventions: Drug: Rivaroxaban 10 MG
- Rivaroxaban 20mg daily (Experimental): orally, 10 mg twice daily for day1 and day 2 after femoral venepuncture
  Interventions: Drug: Rivaroxaban 20 MG
- Low-molecular-weight heparin (Active Comparator): subcutaneously, 0.4 ml once daily, before femoral venepuncture (day1) and after the day of femoral venepuncture (day 2)
  Interventions: Drug: Low-molecular-weight heparin

INTERVENTIONS:
Drug: Rivaroxaban 10 MG — Rivaroxaban pill 10mg qd, day1 and day2 after femoral venepuncture
  Arms: Rivaroxaban 10mg daily
Drug: Rivaroxaban 20 MG — Rivaroxaban pill 10mg bid, day1 and day2 after femoral venepuncture
  Arms: Rivaroxaban 20mg daily
Drug: Low-molecular-weight heparin — 0.4 ml once daily, before femoral venepuncture(day1) and the following day (day 2)
  Arms: Low-molecular-weight heparin

SUMMARY:
The study is designed to compare the efficacy and safety of oral rivaroxaban and subcutaneous low-molecular-weight heparin in preventing femoral venepuncture associated thrombosis among cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85
* Histologically or cytologically confirmed advanced or metastatic solid tumors
* Patients will be received femoral venepuncture for apheresis by cell separator, which is the necessary process to perform following adoptive cell immunotherapy.
* Estimated life expectancy > 3 months
* Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5 (unless patient is receiving warfarin in which case PT-INR must be <3), PTT <1.5X ULN
* Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.

Exclusion Criteria:

* known conditions associated with high risk of bleeding, known history of hemorrhagic diathesis
* Platelet count < 50 000 G/L
* Active bleeding
* Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune related thyroid disease and vitiligo are permitted.
* Patients with obstructive jaundice
* Patients with Spleen hyperfunction
* Presence of an active acute or chronic infection including: a urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Pregnant or breast-feeding women，or lack of effective contraceptive treatment for women of childbearing age.;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of deep venous thrombosis | 4 weeks
  the incidence of deep venous thrombosis of the legs by the systematic examinations performed at the end of the 4-week after femoral venepuncture

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 4 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v 3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical Unvierstiy Cancer Center/ Beijing Shijitan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Wang S, Morse MA, Jiang N, Zhao Y, Song Y, Zhou L, Huang H, Zhou X, Hobeika A, Ren J, Lyerly HK. Prospective randomized comparative study on rivaroxaban and LMWH for prophylaxis of post-apheresis thrombosis in adoptive T cell immunotherapy cancer patients. J Thromb Thrombolysis. 2019 May;47(4):505-511. doi: 10.1007/s11239-019-01844-7. PMID 30903459